CLINICAL TRIAL: NCT02292264
Title: Risk Factors and Complications of Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, Zealand University Hospital
Other Study IDs: HS_01
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical treatment of ventral hernia: Adult patients who underwent a ventral hernia Repair at Zealand University hospital

SUMMARY:
The aim of this study is to evaluate risk factors and complications of ventral hernia repair. A retrospective study of journal files with patients undergoing ventral hernia repair, and an analyses of complications by use of the Clavien-Dindo classification of surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Surgically treated ventral hernia repair

Exclusion Criteria:

* All surgically treated patients are included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent ventral hernia repair at the Surgical Department of Køge University Hospital in the timeperiod from 2009 - 2014.
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Identifying pre-operative risk factors by use of the Clavien Dindo classification. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Sjølander, MS, Principal Investigator — Dept. of surgery, Køge University Hospital
Locations (1):
- Køge University Hospital, Køge, Denmark